CLINICAL TRIAL: NCT06232668
Title: Molecular Study of the Maternal-fetal Interface Prospectively to the Onset of Preeclampsia Using Single Cell Technology.
Brief Title: Molecular Study of the Maternal-fetal Interface in Preeclampsia.
Acronym: PREMAFE
Status: Recruiting | Type: Observational
Sponsor: Carlos Simon Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: FCS-IMF-TG-23-03
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Early onset Preeclampsia (EOPE); First trimester; Chorionic villi; Pregnancy; Molecular study; Decidua; Maternal-fetal interface; Other pregnancy complications; Omic techniques
MeSH Terms: conditions — Pre-Eclampsia | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Maternal-fetal interface biopsy (chorionic villi + decidua) and maternal peripheral blood samples with circulating genetic material (C-RNA/C-DNA) and other biomolecules and cellular component to provide preeclampsia information and other obstetric complications.
  * Maternal-fetal interface tissue (placenta and decidua) and maternal peripheral blood samples containing circulating genetic material (C-RNA/C-DNA) and other biomolecules, and cellular components, to support research on preeclampsia and other obstetric complications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases group: Women recruited between 9 and 15 gestational weeks diagnosed with preeclampsia or other complication at the end of pregnancy.
  Interventions: Procedure: Maternal-fetal interface biopsy and peripheral blood collection in cases group
- Control group: Women recruited between 9 and 15 gestational weeks without diagnosis of preeclampsia or other complication at the end of the pregnancy
  Interventions: Procedure: Maternal-fetal interface biopsy and peripheral blood collection in control group

INTERVENTIONS:
Procedure: Maternal-fetal interface biopsy and peripheral blood collection in cases group — Maternal-fetal interface tissue (chorionic villi and decidua) will be collected from women who have a recommendation for aneuploidy testing, and the remaining fragment will be used for this study and peripheral blood collection in cases group. Clinical data will be compiled.
  Groups: Cases group
Procedure: Maternal-fetal interface biopsy and peripheral blood collection in control group — Maternal-fetal interface tissue (chorionic villi and decidua) will be collected from women who have a recommendation for aneuploidy testing, and the remaining fragment will be used for this study and peripheral blood collection in control group. Clinical data will be compiled.
  Groups: Control group

SUMMARY:
Preeclampsia (PE) is a major obstetric complication with short- and long-term consequences for the mother and the fetus. Early screening tools to reduce its mortality and morbidity, as well as to prevent the life-threatening consequences are needed. Thus, the detection of women at risk of suffering PE is key to apply preventive and treatment strategies. Recently, the maternal contribution to PE based on defective decidualization that prevents the establishment of a functional maternal-fetal interface has been evidenced. The main objective of this study is to identify molecular markers or aberrant maternal-fetal cell types that can be detected early in the development of the disease in maternal-fetal interface tissue (chorionic villi + decidua) collected during gestational weeks 9 to 15. Maternal-fetal interface biopsy will be collected from women who have a recommendation for aneuploidy testing. The remaining fragment will be used for this study.

DETAILED DESCRIPTION:
The hypothesis is that those women who develop PE have impaired decidualization associated with shallow cytotrophoblast invasion during the development of the maternal-fetal interface whose molecular profile analysis at the single cell level will allow characterization of PE development prior to the onset of symptoms.

The purposed study is a biomedical, prospective, multicentre, case-control aimed to characterize the molecular profile of the maternal-foetal interface in the first trimester of pregnancy early in the development of preeclampsia using single-cell sequencing technology. Distinguishing the maternal and fetal origin of the chorionic biopsy cells , describing the maternal-foetal interface and deciphering the intercellular communications and altered pathways in PE and other obstetric complications could be suggested as a secondary outcome, as well as the characterization of the blood sample, the epigenome and metabolome of single cells or the validation of markers of the different cell types. . Another objective will be to perform a molecular characterization of maternal-fetal blood and tissue samples collected at the time of delivery, with the aim of correlating the alterations detected in the first trimester with the molecular profiles at the end of pregnancy in both PE patiens and controls.

Subjects will be 2084 pregnant women over the age of 18 recruited between 9 and 15 gestational weeks. Patients attending the participating referral centers for a chorionic villus biopsy due to the detection of a foetal chromosomal abnormality risk will provide the leftover chorionic biopsy sample after determination of the risk of trisomies and a peripheral blood sample for genotyping of maternal lymphocytes and circulating cRNA.

Data will be registered in an electronic Case Report Form (eCRF) specifically designed for this study. Monitoring activities and data verification will be performed during the whole study to ensure data quality, integrity and transparency.

The total estimated duration of the study is 52 months, of which the first 48 months will correspond to the recruitment period of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose written informed consent approved by the Ethics Committee (EC) has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
* Women over the age of 18 at the time of signing the informed consent form.
* Pregnant women with a single gestation between weeks 9 and 15 of gestation who will undergo a chorionic villus biopsy according to the centre's usual clinical practice.

Exclusion Criteria:

* Women with multiple pregnancy.
* Non-evolving pregnancies (including delayed abortion/foetal orbit).

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women over 18 years old
Study Population: Pregnant women over the age of 18 recruited between 9 and 15 gestational weeks who attend the participating referral centers for a chorionic villus biopsy due to the detection of a foetal chromosomal abnormality risk.
Sampling Method: Non-Probability Sample
Enrollment: 2084 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To charactize the molecular profile of the maternal-fetal interface between 9 and 15 weeks of gestation in healthy and preeclamptic pregnancies | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks
  Differentially expressed genes between control vs preeclampsia group at the level of cell types/subtypes

SECONDARY OUTCOMES:
To characterise the molecular profile of the maternal-fetal interface between 9 and 15 weeks of gestation in pregnancies diagnosed with pregnancy complication other than preeclampsia | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks
  Differentially expressed genes between control vs cases group at the level of cell types/subtypes.
To characterize the molecular profile of the maternal-fetal interface at the end of pregnancy in healthy and preeclamptic pregnancies | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks
  Differentially expressed genes between control vs preeclampsia group at the level of cell types/subtypes
To characterise the epigenome and metabolome of individual cells from the maternal-fetal interface in healthy pregnancies and those diagnosed with preeclampsia or other pregnancy complication | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks
  Differentially methylation profiles and differentially metabolites between control vs cases group at the level of cell types/subtypes.
The discovery and validation of molecular markers as candidates for early diagnosis and/or therapy | From the date of enrollment (minimum 9 weeks) until the end of pregnancy (maximum 43 weeks), assessed up to 34 weeks
  Area Under the ROC Curve and/or cell type phenotyping in in vitro cultures after disrupting the candidate

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Garrido, PhD, Principal Investigator — Fundación Carlos Simon para la investigación en salud de la mujer
Locations (5):
- Spain (5):
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante
  - Hospital Universitario de Torrejón, Madrid, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia